CLINICAL TRIAL: NCT01203553
Title: Mesh Implantation for Prophylaxis of Incisional Hernia
Brief Title: Prophylactic Mesh Implantation for the Prevention of Incisional Hernia
Acronym: ProphMesh
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK 094/10
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Incisional Hernias
Keywords: Incisional hernias; Prophylaxis; Preperitoneal mesh
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: The main operation will be performed as planned. For the closure of the abdominal wall, a standard technique will be applied using a running suture of PDS 1 loop. The distance of the sutures to the fascial border is 1cm and the distance between two stitches is not more than 1cm. The total length of suture is at least 4 times the total length of the abdominal incision
  Interventions: Procedure: Abdominal surgery
- Treatment Group: The main operation will be performed as planned. Prior to the closure of the abdominal wall a mesh will be implanted in a standardized fashion: A Dynamesh IPOM mesh will be used for the present study. The mesh has a width of 15cm and is tailored to overlap lateral and cranial boarders at least 5cm. The mesh will be placed intra-abdominally and fixed using intra-abdominal stitches using Prolene 2/0 in all four corners. After the initial fixation of the mesh in all quadrants, the boarders of the mesh will be adapted using Prolene 2/0 running sutures. The fixation aims to prevent any intestinal structures to herniate onto the mesh. Afterwards, the abdominal wall is closed as described in the control group.
  Interventions: Procedure: Abdominal surgery

INTERVENTIONS:
Procedure: Abdominal surgery — Intraoperative mesh implantation

SUMMARY:
Incisional hernias are primarily repaired using prosthetic meshes. In Switzerland such meshes are mainly implanted via open or laparoscopic approach. The differential impact of these two types of surgical technique on recurrence rate will be investigated with this study.

With this multicenter cohort study the outcomes of laparoscopic and open incisional hernia repair will be investigated prospectively. Hernia recurrence is the main outcome measure.

DETAILED DESCRIPTION:
Background

Incisional hernia is one of the most common complication in general abdominal surgery. An overall incidence of 20% has been found in retrospective studies, ranging in up to 50% of patients with selected risk factors such as obesity.

In the general surgical patient the current standard is the closure of the abdominal wall using a running, slowly absorbable suture. With this well established clinical practice the incidence remains high and incisional hernia repair must be performed frequently in order to treat patients'symptoms and to prevent progression of the hernia an possible complications.

Consequently, in high risk patients prophylactic mesh implantation is performed routinely in our institution.

Objective

* Occurrence of at least two of the following factors:

  * Male gender
  * Malignant tumor present
  * Body mass index above 25kg/m2
  * Previous laparotomy
* Elective operation
* Patient >18 years
* Written informed consent

Methods

Prospective,two armed, controlled, randomized study

ELIGIBILITY:
Inclusion Criteria:

* Occurrence of at least two of the following factors:

  * Male gender
  * Malignant tumor present
  * Body mass index above 25
  * Previous laparatomy
* Elective operation
* Patient > 18 years
* Written informed consent

Exclusion Criteria

* Previous intra-abdominal mesh placement
* Emergency procedures
* Previous incisional hernia
* Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with a high risk for incisional hernia formation
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Incidence of incisional hernia | 3 years

SECONDARY OUTCOMES:
Direct in-hospital costs | 3 years
Intraoperative complications | 3 years
Postoperative complications | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Prof. Dr. med., Principal Investigator — Berne, University Hospital, Univesrity of Berne, Switzerland
Locations (1):
- Dep. of Visceral and transplant surgery, Berne University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Kohler A, Lavanchy JL, Lenoir U, Kurmann A, Candinas D, Beldi G. Effectiveness of Prophylactic Intraperitoneal Mesh Implantation for Prevention of Incisional Hernia in Patients Undergoing Open Abdominal Surgery: A Randomized Clinical Trial. JAMA Surg. 2019 Feb 1;154(2):109-115. doi: 10.1001/jamasurg.2018.4221. PMID 30476940